CLINICAL TRIAL: NCT03015441
Title: Evaluation of a 28-day Fermented Milk Product Consumption Twice Daily as Compared to a Non-fermented Milk Product on Intestinal Gas Production in Healthy Subjects High Dihydrogen Producers A Randomized, Controlled, Double-blind, Parallel Arms, Adaptive Study
Brief Title: Evaluation of a 28-day Fermented Milk Product Consumption Twice Daily as Compared to a Non-fermented Milk Product on Intestinal Gas Production in Healthy Subjects High Dihydrogen Producers
Acronym: BREEZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NU378
Record Dates: First submitted 2017-01-02; First posted 2017-01-10 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Excessive Intestinal Gas Production
Keywords: Healthy subjects; Probiotics; Breath test; Dihydrogen; Methane; Intestinal gas production; Gut microbiota

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Fermented milk product containing probiotics (Other)
  Interventions: Other: Milk product fermented by lactic bacteria or not fermented
- Arm 2: Milk-based non-fermented dairy product (Other)
  Interventions: Other: Milk product fermented by lactic bacteria or not fermented

INTERVENTIONS:
Other: Milk product fermented by lactic bacteria or not fermented — 2 pots of 125g consumed daily during 28 days

SUMMARY:
The purpose of this study is to assess the effect of a 28-day fermented milk product consumption twice daily on intestinal gas production of dihydrogen (H2) and methane (CH4) in healthy subjects high H2 producers.

ELIGIBILITY:
Inclusion Criteria:

* Subject with body mass index (BMI) between 18.0 and 30.0 kg/m2 (bounds excluded)
* Subjects having a high dihydrogen (H2) production as defined by a fasting exhaled level of H2 in breath at 10 parts per million (ppm) or more.
* Women of childbearing potential must be using a medically approved method of contraception OR women must be postmenopausal for at least 12 months prior to study entry

Exclusion Criteria:

* Subject with functional gastrointestinal disorder according to ROME III criteria (Functional Bowel Disorders/FBD module, Functional Dyspepsia/FD module, Irritable Bowel Syndrome/IBS module)
* Subject with gastrointestinal disorders according to investigator's medical assessment
* Subject taking drugs that might modify gastrointestinal function
* Subject with severe disease as assessed by the investigator (ex: cancer, severe heart disease, kidney disease, neurological disease or psychiatric disease, immunodeficiency disorder)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2017-05-04 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Comparison between groups of the change from baseline (Day0) of breath H2 production elicited by a lactulose challenge test after 28 days of investigational product consumption | Baseline and after 28 days

SECONDARY OUTCOMES:
Comparison between groups of the change from baseline (Day0) of breath H2 production elicited by a lactulose challenge test after 14 days of investigational product consumption | Baseline and after 14 days
Comparison between groups of the change from baseline (Day0) of breath CH4 production elicited by a lactulose challenge test after 14 days and 28 days of investigational product consumption | Baseline, after 14 days and after 28 days
Comparison between groups of the change from baseline (Day0) in the fasting breath H2 and CH4 values after 14 days and 28 days of investigational product consumption | Baseline, after 14 days and after 28 days

OTHER OUTCOMES:
Comparison between groups of the change in composition and activity of gut microbiota from stool samples collected before and after 28 days of investigational product consumption | Baseline, after 28 days
Adverse event | AE and SAE assessment through study completion and up to 14 days after the last study visit

CONTACTS AND LOCATIONS:
Overall Officials: Boris Le NEVE, PhD, Study Chair — Danone Research, Palaiseau, France
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No